CLINICAL TRIAL: NCT04991623
Title: Short-term Effects Kinesiology Tape on Sitting Postural Control in Moderate and Severe Cerebral Palsy
Acronym: KT-SIT_CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: jma003
Record Dates: First submitted 2021-07-21; First posted 2021-08-05 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy; Kinesiology Taping; Postural Control
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiology taping (Experimental): Apply a kinesiology taping on the abdominal muscles plus conventional physiotherapy
  Interventions: Device: Kinesiology taping
- Physiotherapy Group (Active Comparator): Apply a conventional physiotherapy
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Device: Kinesiology taping — We used kinesiology taping in abdominal muscles
  Arms: Kinesiology taping
Other: Conventional physiotherapy — We used conventional physiotherapy to comparate
  Arms: Physiotherapy Group

SUMMARY:
To analyze the short-term effect of kinesiology taping on sitting postural control in moderate and severe cerebral palsy

ELIGIBILITY:
Inclusion Criteria:

* age between 4 and 14 years
* diagnosis of motor and cognitive disability
* have prescribed physiotherapy treatment at school
* acquisition of autonomous sitting
* sign the consent informed

Exclusion Criteria:

* presentation of an allergic reaction to tape
* presentation of wounds in the area of application of the tape
* having received botulinum toxin treatment in the last 6 months

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Posture and Postural Ability Scale - T0 | pre-intervention
  Posture and Postural Ability Scale pre-intervention (PPAS pre). Score from 0 to 7, and the higher the score, the better posture
Posture and Postural Ability Scale - T1 | at 10 days
  Posture and Postural Ability Scale post-intervention (PPAS post). Score from 0 to 7, and the higher the score, the better posture
Segmental Assessment of Trunk Control - T0 | pre-intervention
  Segmental Assessment of Trunk Control pre-intervention (SATco pre). Score from 1 to 7, and the lower the score, the better balance
Segmental Assessment of Trunk Control - T1 | at 10 days
  Segmental Assessment of Trunk Control post-intervention (SATco post).Score from 1 to 7, and the lower the score, the better balance

CONTACTS AND LOCATIONS:
Overall Officials: Javier Merino Andrés, MSc, Principal Investigator — Researcher
Locations (1):
- Javier Merino Andrés, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No